CLINICAL TRIAL: NCT04329611
Title: A Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of Oral Hydroxychloroquine for the Treatment of SARS-CoV-2 Positive Patients for the Prevention of Severe COVID-19 Disease.
Brief Title: ALBERTA HOPE COVID-19 for the Prevention of Severe COVID19 Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolment was suspended on 22may2020, after Mehra et al (Lancet 2020) then stopped due to lack of Covid19 cases.
Sponsor: Dr. Michael Hill (Other)
Collaborators: Alberta Health services (Other); University of Alberta (Other); University of Calgary (Other); Calgary Health Trust (Other); Alberta Innovates Health Solutions (Other); Government of Alberta (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Michael Hill, Co-Principal Investigator, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ABCOV-01 version 1.5
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: SARS-Cov2; viral pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomization will be conducted using an online tool. The use of an online tool will allow for dynamic randomization which ensures concealment of allocation. We will use a minimal sufficient balance randomization tool to ensure balance on age, sex, risk status (binary variable based on immune competence and other identified risks), days from symptom onset to randomization and provincial health zone (5 categories). These variables will be identified at telephone screening by a study coordinator, clarified with a physician when necessary, and entered into the online randomization tool. It is predicted that many patients will want treatment. Further, immunosuppressed patients may be at the highest risk of fatal outcomes. Therefore, we will use 2:1 randomization (HCQ: placebo).
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomized, double-blind, placebo-controlled trial - trial staff and patients will all be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxychloroquine (Active Comparator): hydroxychloroquine 400 mg po bid loading dose for 1 day followed by 200 mg po twice daily for 4 days
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — COVID19
  Other Names: plaquenil

SUMMARY:
Albertans with COVID-19 are at risk of deteriorating and developing severe illness. Those over age 40 or with co-morbid illness, and likely those who are immune suppressed, are at highest risk. This study will include a focus on people with immune-suppressed states. Individuals confirmed to have SARS-CoV-2 infection will be identified using administrative data (positive lab result, age 18 or over, not hospitalized, and not living in SL4 level of care). They will then be contacted by AHS staff, independent of the researchers, to obtain their consent for the researchers to contact them about this trial. The AHS staff member who contacts the individual will enroll consenting individuals into a study database. If they provided an email address an email will automatically be sent to the individual with study information. Those who decline to be contacted will also be informed of the study website so they can choose to review the study information and self-enrol, although they will need to do so quickly to meet study timelines. Enrolled participants will be contacted by a study coordinator. Those without access to the internet will be informed about the study details when they are contacted by a study coordinator. When the study coordinator contacts potential participants the study will be reviewed, and the potential participant will have an opportunity to ask questions. Consent for participation will be obtained by telephone. Telephone consent will be recorded. Participants will then be screened for inclusion and exclusion criteria by telephone interview and review of Alberta Netcare. Alberta Netcare is the province of Alberta's public Electronic Health Record used to store patient information so that it is easily accessible to healthcare professionals for the purpose of care. Information like immunizations, ECG results, diagnostic images and reports, written medical reports (e.g. surgery reports, consultations, hospital admissions), diagnostic lab testing results (e.g. blood tests, urine tests, blood bank info), allergies and intolerances (drug and food allergies, food intolerances), prescription history, and general patient information (e.g. name, birthdate, personal health number, address, phone number). Those who are not eligible for the study will be informed of the reason(s) for ineligibility (generally it will be a safety exclusion and they should be aware of this). Those who are eligible will be randomized to receive HCQ or placebo for a total duration of 5 days. Study drug will be delivered to their residence by courier. Telephone follow-up will occur at day 7 (range 7-10 days) and at day 30 (range 25-35 days).

DETAILED DESCRIPTION:
This double-blind placebo-controlled, randomized clinical trial will determine if hydroxychloroquine for 5 days, initiated within 96 hours of confirmation of a positive COVID-19 result, and within 12 days of symptom onset, reduces the occurrence of severe COVID-19 disease. Severe disease is defined as the composite of hospitalization, invasive mechanical ventilation and 30-day mortality. This trial will enrol consenting adults who are not hospitalized, are age 18 or over, have a risk factor for severe disease, have no contraindication to treatment with hydroxychloroquine, can swallow pills, and who do not have a severe underlying comorbidity where treatment is not likely to be beneficial to the patient.

Secondary outcomes will be the proportion of participants requiring hospitalization, invasive mechanical ventilation, 30-day mortality, and disposition at 30 days, defined as recovered, ongoing symptoms but not hospitalized, hospitalized, or deceased.

Randomization will be stratified by age, risk of severe disease, and Alberta Health zone of primary residence. A pre-specified risk classification that includes immunosuppressed status will define those at high risk of severe disease. Health care delivery across Alberta Health zones will likely differ, in part due to the remote location of most patients in some zones.

Alberta has a single publicly funded health care system with processes and administrative data that will allow complete capture of health system encounters and resource utilization. The population is ethnically diverse. In 2016, 23.5% of Albertans belonged to a visible minority group compared with 22.3% for Canada overall (1). Also, in 2018, 94.1% of Albertans age 15 and older used the internet for personal use compared with 91.3% for Canada overall; this excluded full-time residents of institutions (2). This will support a high degree of electronic recruitment and data capture.

The current COVID-19 epidemic has also paused most ongoing research, thus providing access to many experienced researchers and highly trained research staff.

Lack of any proven treatments for this severe condition makes it imperative that we use the resources we have to try to improve the lives of Albertans and determine if there is evidence for the use of hydroxychloroquine for confirmed COVID-19 disease, overall, and in high risk participants.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection, defined as RT-PCR provincial laboratory confirmation.
2. Self-reported symptoms of SARS-CoV-2 infection including any of the following: fever ≥37.5°C, cough, dyspnea, chest tightness, malaise, sore throat, myalgias, or coryza
3. Time from a positive test result to day 1 of treatment within 4 days
4. Time from patient reported first symptoms to day 1 of treatment within 12 days
5. Adults, age 18 and over, with any risk factor for severe disease
6. Resident of Alberta or if not a resident of Alberta able to provide complete follow-up data
7. Agrees to use adequate contraception for the duration of the study
8. Informed consent

Exclusion Criteria:

1. Currently or imminently planned admission to hospital
2. Any contraindication to hydroxychloroquine :

   1. Known hypersensitivity to hydroxychloroquine, chloroquine, or other 4-aminoquinoline derivatives, or any component of the formulation
   2. Known diagnosis of G6PD deficiency or porphyria
   3. Known retinal eye disease with vision impairment, in which hydroxychloroquine is a known contraindication
   4. Known history of QTc prolongation or QTc of > 470 msec (males) or > 480 msec (females) on any ECG within the previous year, if available
   5. Unexplained syncope or family history of long QT syndrome or family history of premature sudden cardiac death at < 50 years of age
   6. Severe diarrhea and/or vomiting or any eating disorders or any persistent vomiting condition
   7. Known significant liver disease including cirrhosis associated with any history of ascites, encephalopathy, or variceal bleeding as per history or medical chart (or Child Pugh B&C) or alcoholic hepatitis
   8. Uncontrolled epilepsy (more than 2 seizures within the previous year or any hospitalizations for status epilepticus within the previous 2 years)
   9. Current use of hydroxychloroquine (Plaquenil), chloroquine, lumefantrine, mefloquine, quinine, artemether, cyclosporine, dapsone, digoxin, and drugs that are known to prolong the QTc as per section 7.5.2.
   10. Score of 7 or more on the Tisdale scale modified such that instead of (1) admission potassium, any known serum potassium within the previous 30 days will be used; if no serum potassium is available the sub-score will be 0, and (2) admission ECG, any known ECG within the previous year will be used; if no ECG is available, the sub-score will be 0; (3) Use of HCQ will be included as one risk factor and anyone concurrently using a medication from the list of drugs known to prolong the QTc will already be excluded. (The other major risk factors for prolonged QTc are sepsis, heart failure, acute myocardial infarction, none of which are likely to be encountered in the outpatient setting).
3. Participation in an ongoing interventional clinical trial within the previous 30 days
4. Use of hydroxychloroquine (Plaquenil) or chloroquine, lumefantrine, mefloquine, or quinine within the previous 30 days.
5. Inability to swallow pills or any other reason that compliance with the medical regimen is not likely
6. Pregnant or breastfeeding
7. Severe underlying disease where treatment is not likely to be beneficial to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Composite of hospitalization, invasive mechanical ventilation or death within 30 days | Within 30 days of randomization
  The aim of this intervention is to prevent severe COVID-19 disease.
  This trial aims to confirm that severe COVID-19 disease can be reduced by a relative risk reduction of 50% by the use of hydroxychloroquine.The aim of this intervention is to prevent severe COVID-19 disease.
  This trial aims to confirm that severe COVID-19 disease can be reduced by a relative risk reduction of 50% by the use of hydroxychloroquine.The aim of this intervention is to prevent severe COVID-19 disease.
  This trial aims to confirm that severe COVID-19 disease can be reduced by a relative risk reduction of 50% by the use of hydroxychloroquine.

SECONDARY OUTCOMES:
mortality | Within 30 days of randomization
  Mortality within 30 days of randomization
Symptom duration | Within 30 days of randomization
  defined as the number of days from randomization to complete symptom resolution, based on public health follow-up and day 7 and day 30 telephone interview (continuous)
Disposition at 30 days defined as recovered, ongoing symptoms but not hospitalized, hospitalized, or deceased (categorical) | Within 30 days of randomization
  Disposition of the patient at the Day 30 telephone followup

CONTACTS AND LOCATIONS:
Overall Officials: Luanne Metz, MD, Principal Investigator — University of Calgary; Michael D Hill, MD, Study Director — University of Calgary
Locations (2):
- Canada (2):
  - University of Calgary/Foothills Medical Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 24 months after study close out.
Access Criteria: pending.

REFERENCES:
- [Derived] Ganesh A, Rosentreter RE, Chen Y, Mehta R, McLeod GA, Wan MW, Krett JD, Mahjoub Y, Lee AS, Schwartz IS, Richer LP, Metz LM, Smith EE, Hill MD; Alberta HOPE COVID-19 Collaborators. Patient-reported outcomes of neurologic and neuropsychiatric symptoms in mild COVID-19: a prospective cohort study. CMAJ Open. 2023 Aug 8;11(4):E696-E705. doi: 10.9778/cmajo.20220248. Print 2023 Jul-Aug. PMID 37553227
- [Derived] Schwartz I, Boesen ME, Cerchiaro G, Doram C, Edwards BD, Ganesh A, Greenfield J, Jamieson S, Karnik V, Kenney C, Lim R, Menon BK, Mponponsuo K, Rathwell S, Ryckborst KJ, Stewart B, Yaskina M, Metz L, Richer L, Hill MD; ALBERTA HOPE COVID-19 Collaborators. Assessing the efficacy and safety of hydroxychloroquine as outpatient treatment of COVID-19: a randomized controlled trial. CMAJ Open. 2021 Jun 18;9(2):E693-E702. doi: 10.9778/cmajo.20210069. Print 2021 Apr-Jun. PMID 34145052